CLINICAL TRIAL: NCT00403221
Title: A Phase I Study of In-Situ, Neoadjuvant, Pre-Radical Prostatectomy RTVP-1 Gene Therapy in Patients With Locally Advanced Adenocarcinoma of the Prostate (SPORE)
Brief Title: Phase I - Pre-Radical Prostatectomy RTVP-1 Gene Therapy for Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Dov Kadmon, Professor of Urology, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-11112; P50CA058204 (NIH)
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Prostatic Neoplasms
Keywords: Gene therapy; Prostate cancer; Immunology, Angiogenesis inhibition; Phase I clinical trial
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Genetic: RTVP-1 Gene — Cohort Level #1 1.0 x 1010vp Cohort Level #2 5.0x1010vp Cohort Level #3 1.0 x 1011vp Cohort Level #4 5.0x1011vp Cohort Level #5 1.0 x 1012vp Cohort Level #6 5.0x1012vp
  One dose only followed by a radical prostatectomy 4 weeks later.

SUMMARY:
The purpose of this study is to conduct a Phase I clinical trial involving in situ RTVP-1 gene therapy for prostate cancer. We will conduct necessary safety evaluations on a new adenovirus that contains the human genes for RTVP-1. This virus will then be evaluated for safety in men with prostate cancer prior to radical prostatectomy. Based on the preclinical data, we hope that this treatment will induce not only a local cytotoxic and antiangiogenic effect but also, a systemic antitumor immune response capable of eradicating micrometastatic disease (the reason for recurrence in many of these patients).

DETAILED DESCRIPTION:
The population selected for this study includes patients with locally advanced and/or poorly differentiated tumors. These patients have an unacceptably high failure rate when treated by radical prostatectomy alone (over 50% fail within 5 years). The pattern of failure varies. While some patients present with a local recurrence, many have both a local recurrence and distant metastases, or just distant metastases. It is reasonable to assume that many, if not most of these patients, actually harbor micrometastases, present but undiagnosed clinically, at the time of their radical prostatectomy. Our hypothesis is that the cytotoxic, proapoptotic, antiangiogenic and immune stimulatory activities of in-situ RTVP-1 gene therapy will lower the incidence of local tumor recurrences when given to patients prior to surgery. The second part of our hypothesis is that RTVP-1 gene therapy will induce a systemic anti-tumor immune response, which will eliminate pre-existing micrometastases in some of these patients and lower the overall failure rate.

While this Phase I study is not designed to answer these questions, we hope to obtain mechanistic evidence in support of this hypothesis. A Phase II study will then be proposed (and properly powered), to study the efficacy of this approach.

Based on our experience with HSV-tk and GCV in-situ gene therapy, it appears that maximal immune stimulation occurs about 2 weeks following vector injection. Furthermore, repeat injections of an adenoviral vector do not result in excess toxicity or in the generation of anti-adenoviral antibodies sufficient to suppress vector activity. We propose here an intraprostatic injection of RTVP-1 in an adenoviral vector 4-6 weeks prior to radical prostatectomy, in order to allow full expression of the gene therapy tissue effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of prostatic adenocarcinoma without evidence of regional and/or distant metastasis, clinical stage T1c, T2 or T3 with high grade disease (Gleason's 7 - 10) on initial biopsy, or PSA greater than 10 ng/ml with any stage or Gleason score.
* Recent (equal to or less than 1 month prior to study entry) negative bone scan and CT scan of abdomen/pelvis.
* Life expectancy of at least 10 years.
* Appropriate surgical candidate for radical prostatectomy and a performance status of equal to or less than 2 (Zubrod scale).
* Patients should have adequate bone marrow function defined as an absolute peripheral granulocyte count equal to or greater than 1,500 and platelet count of equal to or greater than 100,000, adequate hepatic function with a bilirubin equal to or less than 1.5 mg per cent and SGPT less than 2 x the upper limits of normal, adequate renal function defined as serum creatinine equal to or less than 2.0 mg per cent.
* Patients must have normal coagulation profile (PT, PTT) and no history of substantial non-iatrogenic bleeding diatheses. Use of anticoagulants is limited to local use only (for control of central line patency).
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with the policies of the institution.

Exclusion Criteria:

* Previous or current hormonal treatment, chemotherapy, radiation therapy, immunotherapy or other investigational status drug within the past 4 weeks.
* Unable to tolerate transrectal ultrasound.
* Patients who are not appropriate surgical candidates for radical prostatectomy based on the evaluation of co-existent medical diseases and competing causes of death.
* Patients with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorders are not eligible.
* Patients who are HIV positive or have chronic hepatitis B or C infections are not eligible (because of possible immune effects of these conditions).
* Patients with a history of primary or secondary immunodeficiency or patients taking immunosuppressive drugs such as corticosteroids continuously for greater than 4 months [greater than 5 mg hydrocortisone/day] are ineligible. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have a decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Assessment of safety/toxicity | After treatment with 3-6 patients per cohort level, the patients will be assessed for the frequency of complications to be assured that they do not exceed those anticipated.

SECONDARY OUTCOMES:
To collect data on the morphologic and cytotoxic changes in the radical prostatectomy specimen | Tumor response as measured by cytoreduction is not likely to be the major effect of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dov Kadmon, M.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine - Scott Department of Urology, Houston, Texas, United States

REFERENCES:
- [Background] Satoh T, Timme TL, Saika T, Ebara S, Yang G, Wang J, Ren C, Kusaka N, Mouraviev V, Thompson TC. Adenoviral vector-mediated mRTVP-1 gene therapy for prostate cancer. Hum Gene Ther. 2003 Jan 20;14(2):91-101. doi: 10.1089/104303403321070793. PMID 12614561
- [Background] Ren C, Li L, Goltsov AA, Timme TL, Tahir SA, Wang J, Garza L, Chinault AC, Thompson TC. mRTVP-1, a novel p53 target gene with proapoptotic activities. Mol Cell Biol. 2002 May;22(10):3345-57. doi: 10.1128/MCB.22.10.3345-3357.2002. PMID 11971968
- [Background] Ren C, Li L, Yang G, Timme TL, Goltsov A, Ren C, Ji X, Addai J, Luo H, Ittmann MM, Thompson TC. RTVP-1, a tumor suppressor inactivated by methylation in prostate cancer. Cancer Res. 2004 Feb 1;64(3):969-76. doi: 10.1158/0008-5472.can-03-2592. PMID 14871827
- [Background] Naruishi K, Timme TL, Kusaka N, Fujita T, Yang G, Goltsov A, Satoh T, Ji X, Tian W, Abdelfattah E, Men T, Watanabe M, Tabata K, Thompson TC. Adenoviral vector-mediated RTVP-1 gene-modified tumor cell-based vaccine suppresses the development of experimental prostate cancer. Cancer Gene Ther. 2006 Jul;13(7):658-63. doi: 10.1038/sj.cgt.7700919. Epub 2006 Feb 17. PMID 16485011
- [Background] Ren C, Ren CH, Li L, Goltsov AA, Thompson TC. Identification and characterization of RTVP1/GLIPR1-like genes, a novel p53 target gene cluster. Genomics. 2006 Aug;88(2):163-72. doi: 10.1016/j.ygeno.2006.03.021. Epub 2006 May 22. PMID 16714093
- See also: Scott Department of Urology Clinical Trials — http://www.baylorurology.org